CLINICAL TRIAL: NCT06925503
Title: Effectiveness of a Mind-Body Conditioning Course for the Management of Physical and Emotional Stressors in University Dance Students
Brief Title: Mind-Body Conditioning Course for University Dance Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Beth Steinberg, Associate Director of Research, Ohio State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024B0224
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-09

CONDITIONS: Perceived Stress; Student Burnout; Resilience; Musculoskeletal Injury; Musculoskeletal Abnormalities
MeSH Terms: conditions — Burnout, Psychological; Musculoskeletal Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Second Year Dance majors (Experimental): Second year Dance majors at The Ohio State University who are enrolled in the required Dance 2802 Seminar/Mind-Body Conditioning course
  Interventions: Behavioral: Mind-Body Conditioning Course
- Third Year Dance majors (No Intervention): The Third Year Dance majors completed Dance 2802 the previous year and did not receive the Mind-Body Conditioning course

INTERVENTIONS:
Behavioral: Mind-Body Conditioning Course — Evidence-based mindfulness intervention curated to the physical and emotional needs of University Dance students
  Arms: Second Year Dance majors

SUMMARY:
Mindfulness in Motion (MIM) is an eight-week evidenced based program designed specifically to help participants learn practical stress reduction, burnout and resiliency building techniques. Content includes didactic instruction, community-building group discussion, mindfulness practices, and gentle yoga. Weekly themes include Willingness to Daily Practice, Mindful Sleep, Vision of Self, Supported by the Breath, Mindful Eating and Yoga, Movement Through Balance, Awareness of Sensation, Clarity and Release, and Staying Grounded and Moving Forward. An Ohio State University endorsed, ADA compliant companion smartphone app reinforces weekly content and offers a variety of individual mind-body and mediations practices.

The evidence-based MIM content has been tailored to meet the physical, mental, and emotional needs of student Dance majors at The Ohio State University and integrated into the Dance 2802 course content as Mind-Body Conditioning for second year students. Over the course of the second year student's fall semester, this study will evaluate the effectiveness of this integrated course content on students' perceived stress, burnout, resilience, musculoskeletal injury and discomfort, and weekly respiratory rates. After the semester long course is completed, the students will also assess how well the Mind-Body Conditioning course content was integrated into the required first year seminar for University Dance majors.

DETAILED DESCRIPTION:
Physical injuries and mental health issues are common in collegiate dance students. Distinct from other college students and student athletes, collegiate dancers must manage required academic courses with regular rehearsals, technique classes, and evaluative performances. The need for adequate sleep, proper nutrition, and physical and mental recovery, often disregarded by dance students, can lead to increased physical injuries, as well as increased stress, burnout, and performance anxiety. While dance tradition is slowly shifting, a focus on perfection relative to body appearance and type, personality, and performance continues to be encouraged and emulated. This focus only serves to exacerbate mental health concerns such as eating disorders, body dissatisfaction, anxiety and depression, that are common in dancers.

Mindfulness-based approaches, including breath practices, progressive relaxation, yoga, and meditation, have shown promise in managing the stress and anxiety of college students including student athletes and those who major in performing arts. These interventions can be implemented as a group class, integrated into course content, or as individual, brief practices available or reinforced through a smartphone app. The Department of Dance at The Ohio State University currently offers Dance 5175/2175, Yoga Theory and Practice, through which students become familiar with the benefits of yoga through a rigorous asana (postures) and pranayama (breathwork) training. This new course, Body-Mind Conditioning for Dancers, will include studio work in mind-body practices, as well as education in the research surrounding the efficacy of mindfulness based interventions for conditioning dancers to their peak performance.

Through a collaboration between The Ohio State University Center for Integrative Health and The Ohio State University Department of Dance, the purpose of this study is to evaluate the effects of integrating an evidence based, eight week mindfulness-based intervention into the OSU Dance 2802 curriculum on student perceived stress, burnout, resilience, physical pain and injury and assess the feasibility of integrating the mindfulness-based intervention into the Dance 2802, Introductory Dance Seminar for second year OSU Dance majors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ability to understand and read English
* Second year OSU Dance majors enrolled in Dance 2802 for Fall 2025 semester
* Third year OSU Dance majors who completed Dance 2802 during the 2024-2025 academic year.
* Access to personal smartphone, either iOS or Android, with sufficient memory to install the Mindfulness in Motion smartphone app, and WiFi (OSU eduroam while in class or on campus and LTE or personal WiFi off campus)

Exclusion Criteria:

* OSU student with a minor in Dance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress | Baseline and on completion of the 8-week intervention
  Perceived Stress Scale-10 (PSS-10). A 10-item self-report measure of perceived stress. It is a measure of the degree to which situations in one's life are appraised as stressful over the past month. The 4-point Likert Scale includes responses of 0 (never), 1 (almost never), 2 (sometimes), 3 (fairly often), and 4 (very often). Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Maslach Burnout Inventory-Students - MBI-GS (S) | Baseline and on the completion of the 8-week intervention
  The MBI-GS (S) is a self-report assessment of perceptions of burnout specific to University students. The 16-items describe students' feelings related to their experiences in the academic setting and encompasses how they view their studies and reactions to their academic work. Three sub scales measure exhaustion, cynicism, and professional efficacy. The Likert Scale responses include 0 (never), 1 (a few times a year or less), 2 (once a month or less), 3 (a few times a month), 4 (once a week), 5 (a few times a week), and 6 (every day). The sub scale score for exhaustion can range from 0 to 30 with higher scores indicating higher levels of exhaustion. The sub scale score for cynicism can range from 0 to 30 with higher scores indicating higher levels of cynicism. The sub scale score for professional efficacy can range from 0 to 36 with higher scores indicating increased professional efficacy.
Resilience | Baseline and on completion of the 8-week intervention
  The Connor-Davidson Resilience Scale-10 (CD-RISC-10) is a 10 item self-report assessment of a person's ability to bounce back after adversity. A 5-point Likert Scale for each statement ranges from 0 (not true at all), 1 (rarely true), 2 (sometimes true), 3 (often true), 4 (true nearly all of the time). A respondent's total score can range from 0 to 40 with higher scores indicating higher resilience.
Respiratory Rate | The 30-second count of inhalations will be completed by the participant before and after participating in each weekly Mind-Body Conditioning course session over eight weeks.
  A self-measured count of inhalations (respiratory rate) taken over a 30-second time period. The participant will place their right hand over their left chest and count inhalations for a 30-second time period before and after they participate in the Mind-Body Conditioning course at each 8-week session.
Modified Nordic Questionnaire | Baseline and on completion of the 8-week intervention
  The Modified Nordic Questionnaire (mNMQ) is a 14-item scale measuring musculoskeletal discomfort and injury. Question 1 asks the participant to state if they have experienced pain, discomfort, burning, numbness, tingling or other trouble over the past 30 days in their neck, shoulder, elbow/forearm, wrist/hand, upper and lower back, and legs/feet. Questions 2 - 10 asks about the intensity and length of the the pain, discomfort, etc, in any of the body areas noted in Question 1, as well as if the issues have caused issues with normal activities, to see a health care provider, lost time from work/school. Question 11 requests information related to any musculoskeletal or traumatic injuries diagnosed by a health care provider. Questions 12 and 13 request information on headaches experienced by participants and question 14 asks about other health issues including arthritis, thyroid problems, diabetes, lupus, and other autoimmune disorders.

SECONDARY OUTCOMES:
Feasibility of Intervention Measure | Participants will complete after the completion of the 8-week intervention.
  The Feasibility of Intervention Measure (FIM) is a 4-item self-report assessment to evaluate integration of the Mind-Body Conditioning Course into the Dance 2802 curriculum for the University Dance major. Each statement is scored with a 5-point Likert Scale that includes 1 (completely disagree), 2 (disagree), 3 (neither agree nor disagree), 4 (agree), and 5 (completely agree). Total scores range from 4-20 with higher total scores indicating higher feasibility.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that will be shared will include de-identified descriptive data for both the intervention and control groups, including gender, educational level, and mean age. Feasibility of integrating the intervention into the required course content by the intervention group will also be included. Differences in mean scores between intervention and control groups for perceived stress, burnout, resilience, and respiratory rates (pre- and post-intervention) will be shared. Descriptive data for any differences in the modified Nordic Questionnare pre- and post-intervention will be shared.
Supporting Information: ICF, CSR, Analytic Code
Time Frame: 7-30-26 to indefinitely
Access Criteria: De-identified and curated demographic, statistical data, study overview, study consent will be accessible to academic researchers and educators through a data accessibility link once the data to a repository is finalized.